CLINICAL TRIAL: NCT06349187
Title: Association Between Doctor's Digital Competencies and the Level of Emotional Intelligence and Burnout
Brief Title: Digital Literacy and Emotional Intelligence and Professional Burnout Among Doctors
Status: Recruiting | Type: Observational
Sponsor: Limited Liability Company "Docstarclub" (Other)
Responsible Party: Sponsor
Other Study IDs: dsc002
Record Dates: First submitted 2024-03-31; First posted 2024-04-05 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-03

CONDITIONS: Digital Competences; Emotional Intelligence; Emotional Burnout; Doctor Patient Relation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Doctors of various clinical specialties who are currently working in medical field: Participants over the age of 18, with higher medical education, capable
  Interventions: Diagnostic Test: Interview

INTERVENTIONS:
Diagnostic Test: Interview — Interviewing with using the Hall Emotional Intelligence test, the Maslach emotional burnout test, and the test for determining general and specialized digital competencies

SUMMARY:
The role of digital technologies in healthcare is growing. Therefore, the roles and responsibilities of medical professionals are constantly changing and there is a need for continuous professional development. However, according to some authors, today's generation of doctors can be considered as "digital aborigines" [Aungst, Patel, 2020]. Low literacy in the field of e-health has become a major obstacle to digital transformation in developed countries, so digital skills training for healthcare professionals has gradually been introduced in the USA [Adler-Milstein, et al., 2014], Europe [Schreiweis, et al., 2019], Australia [Evolution of eHealth in Australia, 2016].

However, in our opinion, the digital competence of a doctor is not only the ability to work at a computer and use software. The successful development of the digital world is preceded by some psychological and emotional processes.

Computerization and automation of the healthcare system began relatively recently, traditional (paper) document management in medicine is familiar to everyone, but not optimal from the point of view of system management. Therefore, universal digitalization is perceived as something artificially imposed, increasing the workload of doctors, distracting from their main work and shifting the focus from truly therapeutic activities to filling out documentation. As a result, doctors have a range of negative emotions: fear, annoyance, anxiety, despondency, refusal of further contacts, etc., which lead to an aggravation of emotional burnout. The ability to recognize and live through these states, to come to an inner balance, to accumulate an internal resource for further development of new technologies - all this is possible under the condition of the development of emotional intelligence. By developing so-called soft skills, the doctor will be emotionally stable, capable of further advancement and learning new skills, and will easily cope with temporary difficulties and setbacks.

And the final stage, having gained the opportunity to overcome internal obstacles, the doctor is ready to begin mastering specialized digital skills directly related to medical activities: work in medical information systems, remote monitoring, artificial intelligence, medical decision support systems.

The result of the development of a doctor within this model will be not only digital literacy, but also the development of an internally stable personality that easily overcomes any obstacles not only in training, but also in communication with patients and colleagues.

ELIGIBILITY:
Inclusion Criteria:

* respondent has higher medical education
* he is an employee of the any medical department at this moment

Exclusion Criteria:

* There is no higher medical education
* Does not work in medicine at this moment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will conduct a survey among doctors of various specialties who currently work in healthcare institutions
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2024-06-10 (Estimated); Study Completion 2024-06-10 (Estimated)

PRIMARY OUTCOMES:
Completing the survey | 1 month
  The answer to 100% of the interview questions

CONTACTS AND LOCATIONS:
Overall Officials: Anna N. Korobeynikova, Principal Investigator — Limited Liability Company "Docstarclub"
Locations (1):
- Alexandra Demkina, Moscow, Russia